CLINICAL TRIAL: NCT05798767
Title: Preoperative Cognitive Impairment Predicts Postoperative Delirium in Elderly Patients Undergoing General Anesthesia
Brief Title: Preoperative Cognitive Impairment Predicts Postoperative Delirium
Status: Completed | Type: Observational
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PCI and POD
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-01

CONDITIONS: Delirium in Old Age; Neurocognitive Disorders; Cognitive Impairment
MeSH Terms: conditions — Neurocognitive Disorders; Cognitive Dysfunction | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCI group: Patients with a Mini-Cog score of 3 or less were in the PCI group
  Interventions: Behavioral: Neuropsychological tests
- Normal group: Patients with a Mini-Cog score of 3 or 4 were in the normal group
  Interventions: Behavioral: Neuropsychological tests

INTERVENTIONS:
Behavioral: Neuropsychological tests — Cognitive function screening (Mini-Cog; the Mini-mental State Examination, MMSE), depression screening (Patient Health Questionnaire-9, PHQ-9), sleep quality assessment (Pittsburgh Sleep Quality Index, PSQI), and pain assessment (Numeric Rating Scale, NRS) were performed the day before surgery.
  The Short Confusion Assessment Method (CAM) was administered once per day on postoperative days 1 to 5 to evaluate delirium.

SUMMARY:
Preoperative cognitive impairment (PCI) may increase the incidence of postoperative delirium (POD), yet screening for cognitive impairment is rarely performed. This study hypothesized that Mini-Cog for preoperative cognitive impairment screening predicts postoperative delirium. Elderly patients (65 years or older) attending Henan Provincial People's Hospital during the trial period who required elective thoracic surgery were recruited into the study.

DETAILED DESCRIPTION:
We collected data points on demographics and hospital episodes through the electronic medical record the day before surgery. Cognitive function screening (Mini-Cog; the Mini-mental State Examination, MMSE), depression screening (Patient Health Questionnaire-9, PHQ-9), sleep quality assessment (Pittsburgh Sleep Quality Index, PSQI), and pain assessment (Numeric Rating Scale, NRS) were performed, and the time spent on Mini-Cog test and MMSE assessment was recorded. The Short Confusion Assessment Method (CAM) was administered once per day on postoperative days 1 to 5 to evaluate delirium.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years of age or older,
2. elective thoracic surgery,
3. under general anesthesia.

Exclusion Criteria:

1. history of psychiatric disorders,
2. use of any antipsychotic drugs,
3. ASA score >3
4. severe visual, hearing, or physical dysfunction unable to complete the scale
5. advanced malignant tumors of the chest with distant metastases to bone, liver, etc.,
6. history of general anesthesia surgery in the last six months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients attending Henan Provincial People's Hospital during the trial period who required elective thoracic surgery
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
delirium | February 2022 to March 2023
  postoperative delirium accessed by the Short Confusion Assessment Method (CAM)

CONTACTS AND LOCATIONS:
Locations (1):
- Henan People's Hospital, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li F, Miao M, Li N, Zhou J, Sun M, Zhang J. Prevalence of preoperative cognitive impairment among elderly thoracic surgery patients and association with postoperative delirium: a prospective observational study. Front Hum Neurosci. 2023 Jul 20;17:1234018. doi: 10.3389/fnhum.2023.1234018. eCollection 2023. PMID 37545595